CLINICAL TRIAL: NCT04875390
Title: Evaluation of the Effect of Ultrasonographic Guided Erector Spina Plan Block Application on Postoperative Analgesia in Infants Undergoing Laparotomy
Brief Title: Erector Spina Plane (ESP) Block in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ESP
Record Dates: First submitted 2021-05-01; First posted 2021-05-06 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Acute Postoperative Pain
Keywords: erector spina plane block; pediatric patient
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group E (Other): Intraoperative Erector spina plane block ( 0.3 ml/kg bupivacaine 0.25% at thoracic level 7 and 0.3 ml/kg bupivacaine 0.25% bupivacaine at thoracic level 11, totaling 0.6 ml/kg of 0.25% bupivacaine) will be performed after the surgery is completed.
  Interventions: Other: Erector spina plane block
- group L (Other): Intraoperative local infiltration (0.6 ml/kg of 0.25% bupivacaine will be given to the wound lips at the end of the surgery.
  Interventions: Other: local infiltration

INTERVENTIONS:
Other: Erector spina plane block — After the surgery is completed, intraoperative Erector spina plane block will be performed
  Arms: group E
Other: local infiltration — After the surgery is completed, intraoperative local infiltration will be performed
  Arms: group L

SUMMARY:
In this study, we aimed to evaluate the erector spina plane (ESP) block method that we used in our clinic with ultrasonography in pediatric cases between 1 month and 2 years of age who underwent laparotomy.

DETAILED DESCRIPTION:
36 patients who will undergo laparotomy between the ages of 1 month and 2 years in ASA ( American Society of Anesthesiologists) I-II class will be included in the study. patients will be divided into 2 groups. Intraoperative erector spina plane block will be applied to the 1st group (group E) and intraoperative local anesthetic infiltration will be applied to the 2nd group (group L). Postoperative pain will be evaluated with the FLACC (face, legs, activity, crying, consolation) scale.

ELIGIBILITY:
Inclusion Criteria:

* 1 month and 2 years of age
* ASA (American Society of Anesthesiologists) I-II class
* Patients who underwent nephrectomy, pyeloplasty, adrenal tumor excision with unilateral paramedian incision

Exclusion Criteria:

* Patients who underwent laparotomy with a midline incision
* Local infection at the injection site,
* Anatomical anomalies
* Allergies to local anesthetics,
* Coagulopathy,
* Liver, kidney failure patients

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
the 6th hour pediatric pain scale, face ,legs , activity; cry;consolability (FLACC) | 6th hour
  FLACC : Each of the five categories (F)face; (L)legs; (A)activity; (C)cry; (C)consolability is scored from 0-2 which results in a total score between 0 and 10. 0:relaxed and comfortable, 1-3: mild discomfortable, 4-6: moderate pain, 7-10: severe pain

SECONDARY OUTCOMES:
paracetamol consumption | 24 hours
  the total number of paracetamol requirements in the first 24 hours in all patients

CONTACTS AND LOCATIONS:
Overall Officials: Hülya Kaşıkara, Principal Investigator — Ankara City Hospital Bilkent; Sengül Özmert, Study Director — Ankara City Hospital Bilkent; Feyza Sever, Study Director — Ankara City Hospital Bilkent; Halil Kara, Study Director — Yıldırım Beyazıt University Medical Pharmacology
Locations (1):
- hülya KAŞIKARA, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mostafa SF, Abdelghany MS, Abdelraheem TM, Abu Elyazed MM. Ultrasound-guided erector spinae plane block for postoperative analgesia in pediatric patients undergoing splenectomy: A prospective randomized controlled trial. Paediatr Anaesth. 2019 Dec;29(12):1201-1207. doi: 10.1111/pan.13758. Epub 2019 Nov 8. PMID 31630465
- [Background] Aksu C, Sen MC, Akay MA, Baydemir C, Gurkan Y. Erector Spinae Plane Block vs Quadratus Lumborum Block for pediatric lower abdominal surgery: A double blinded, prospective, and randomized trial. J Clin Anesth. 2019 Nov;57:24-28. doi: 10.1016/j.jclinane.2019.03.006. Epub 2019 Mar 6. PMID 30851499